CLINICAL TRIAL: NCT02609724
Title: Effectiveness of Fluoroscopy-guided Manual Lymph Drainage (MLD) Versus Traditional MLD or Placebo MLD, as Part of Decongestive Lymphatic Therapy, for the Treatment of Breast Cancer-related Lymphoedema (BCRL): a Randomised Controlled Trial
Brief Title: Effectiveness of Fluoroscopy-guided MLD for Treatment of BCRL
Acronym: EFforT-BCRL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IWT150178
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Results first posted 2022-03-07 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Breast Neoplasm; Lymphedema
Keywords: breast cancer; lymphedema; manual lymph drainage; near infrared fluorescence imaging
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Skin Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluoroscopy-guided MLD (Experimental): Information, skin care, compression therapy, exercises and fluoroscopy-guided MLD 3 weeks (14 sessions of 60 minutes) of intensive treatment 6 months (18 sessions of 60 minutes) of maintenance treatment 6 months of follow-up
  Interventions: Other: Information; Other: Skin care; Other: Compression therapy; Other: Fluoroscopy-guided MLD
- Traditional MLD (Active Comparator): Information, skin care, compression therapy, exercises and traditional MLD 3 weeks (14 sessions of 60 minutes) of intensive treatment 6 months (18 sessions of 60 minutes) of maintenance treatment 6 months of follow-up
  Interventions: Other: Information; Other: Skin care; Other: Compression therapy; Other: Traditional MLD
- Placebo MLD (Placebo Comparator): Information, skin care, compression therapy, exercises and placebo MLD 3 weeks (14 sessions of 60 minutes) of intensive treatment 6 months (18 sessions of 60 minutes) of maintenance treatment 6 months of follow-up
  Interventions: Other: Information; Other: Skin care; Other: Compression therapy; Other: Placebo MLD

INTERVENTIONS:
Other: Information — During intensive phase: a leaflet with information about the lymphatic system and lymphoedema, clinical evaluation and conservative treatment of lymphoedema During maintenance phase: two informational sessions about self-management and about compression sleeves and other compression material
Other: Skin care — The skin is hydrated during the session. If wounds are present, the wound is cared.
Other: Compression therapy — During intensive phase: application of multi-layer, multi-component bandages During maintenance phase: wearing custom-made compression garment
Other: Fluoroscopy-guided MLD — Fluoroscopy-guided MLD is applied on patient-specific lymphatic system (known from lymphofluoroscopy) by applying cleaning techniques on lymph nodes, resorption techniques to stimulate resorption of lymph by lymph capillaries and gliding technique to stimulate transport of lymph through lymph collectors
  Arms: Fluoroscopy-guided MLD
Other: Traditional MLD — Traditional MLD is applied without knowledge of the patient-specific lymphatic architecture. During MLD no cream or oil is used. A pressure with the hands up to 40 mmHg is applied. Drainage is performed at the level of the jugular and occipital region and the belly (in the depth). Draining techniques are applied on the retroclavicular lymph nodes, axillary lymph nodes, humeral lymph nodes and cubital lymph nodes. At the level of the hand, arm, shoulder and trunk, hand movements are applied to stimulate lymphatic transport through the lymph collectors. The therapist's hands perform 'pumping-movements' while stretching the skin.
  Arms: Traditional MLD
Other: Placebo MLD — During placebo MLD a superficial massage with massage cream is performed on the patient's contralateral arm and on the belly.
  Arms: Placebo MLD

SUMMARY:
The main scientific objective of this multicentric double-blinded randomised controlled trial entails examining the effectiveness of fluoroscopy-guided MLD versus traditional MLD versus placebo MLD, applied as part of the intensive and maintenance phase of Decongestive Lymphatic Therapy, for the treatment of BCRL Secondary scientific objectives entail examining the relationship between different variables of lymphoedema at baseline

DETAILED DESCRIPTION:
According to the International Society of Lymphology, lymphoedema needs to be treated with Decongestive Lymphatic Therapy (Consensus Document ISL 2013). This is a two-stage treatment programme. During the first or intensive phase, lymphoedema has to be maximally reduced. This phase consists of skin care, manual lymph drainage (MLD), multi-layer bandaging and exercise therapy. The second or maintenance phase aims to conserve and optimise the results obtained in the first phase. It consists of skin care, compression by a low-stretch elastic sleeve, exercises and lymph drainage. Skin care, multi-layer bandaging, elastic sleeve and exercises are treatment modalities that (after instructing the patient) can be performed by the patient herself. MLD has to be applied by a physical therapist and hence entails a big financial cost for the patient and the Health Care (Kärki et al 2009). The effectiveness of MLD applied during the intensive phase has been investigated by 5 randomised controlled trials, but there is conflicting evidence. So, further investigation is warranted to determine the relative benefit of MLD. The effectiveness of MLD applied during the maintenance phase has never been investigated (Devoogdt et al 2010, Oremus et al 2012, Huang et al 2013, Ezzo et al 2015).

A possible explanation why MLD is not obviously proven to be effective, is that MLD is applied in an inefficient way: during MLD, hand manoeuvres are applied on all lymph nodes and lymphatics that may be anatomically present. After axillary dissection and/ or radiotherapy (for the treatment of breast cancer), the lymphatic system is damaged: lymph nodes are removed and often fibrosis of the superficial lymphatic system occurs. As a result, rerouting of the lymphatic drainage occurs. Rerouting is patient-specific, consequently, it is possible that the traditional MLD needs be abandoned and a tailored approach needs to be established. Lymphofluoroscopy can aid to apply a more efficient MLD. During lymphofluoroscopy, a fluorescent substance is injected subcutaneously in the hand and it visualizes the transport of lymph from the hand up to the axilla and it demonstrates alternative pathways towards other lymph nodes.

A second explanation why the traditional method of MLD is not proven to be effective, is that research has shown that MLD with high pressure (vs low pressure) is more effective to improve lymph transport, as well as gliding (vs no gliding). During the new method of MLD (or fluoroscopy-guided MLD), the therapist only performs hand movements on functional lymphatics and lymph nodes. In addition, the hand movements are applied with higher pressure and lymph transport through the lymph collaterals is stimulated by applying strikes across the skin.

Therefore, the main scientific objective entails examining the effectiveness of fluoroscopy-guided MLD versus traditional MLD versus placebo MLD, applied as part of the intensive and maintenance phase of Decongestive Lymphatic Therapy, for the treatment of BCRL

ELIGIBILITY:
Inclusion Criteria:

* Age >18y (since the treatment with MLD and the investigation using ICG is not dangerous for pregnant women, women with child bearing age are included)
* Women/ men with breast cancer-related lymphoedema
* Chronic lymphoedema (>3 months present), stage I to IIb
* At least 5% difference between both arms and/ or hands, adjusted for dominance
* Written informed consent obtained

Exclusion Criteria:

* Allergy for iodine, sodiumiodine, ICG
* Increased activity of the thyroid gland; benign tumors of the thyroid gland
* Age <18y
* Oedema of the upper limb from other causes
* Active metastasis of the cancer
* Surgery of the lymphatic system in the past (lymph node transplantation, lymphovenous shunt)
* Cannot participate during the entire study period
* Mentally or physically unable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nele Devoogdt, PhD, Principal Investigator — University of Leuven - KU Leuven and University Hospitals Leuven
Locations (3):
- Belgium (3):
  - Antwerp University Hospital, Antwerp
  - Centre Hospitalier Universitaire (CHU) Sint-Pieter, Lymphoedema Clinic, Brussels
  - University Hospitals of Leuven, lymphovenous center, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang TW, Tseng SH, Lin CC, Bai CH, Chen CS, Hung CS, Wu CH, Tam KW. Effects of manual lymphatic drainage on breast cancer-related lymphedema: a systematic review and meta-analysis of randomized controlled trials. World J Surg Oncol. 2013 Jan 24;11:15. doi: 10.1186/1477-7819-11-15. PMID 23347817
- [Background] Ezzo J, Manheimer E, McNeely ML, Howell DM, Weiss R, Johansson KI, Bao T, Bily L, Tuppo CM, Williams AF, Karadibak D. Manual lymphatic drainage for lymphedema following breast cancer treatment. Cochrane Database Syst Rev. 2015 May 21;2015(5):CD003475. doi: 10.1002/14651858.CD003475.pub2. PMID 25994425
- [Background] Devoogdt N, Christiaens MR, Geraerts I, Truijen S, Smeets A, Leunen K, Neven P, Van Kampen M. Effect of manual lymph drainage in addition to guidelines and exercise therapy on arm lymphoedema related to breast cancer: randomised controlled trial. BMJ. 2011 Sep 1;343:d5326. doi: 10.1136/bmj.d5326. PMID 21885537
- [Background] Devoogdt N, Van Kampen M, Geraerts I, Coremans T, Christiaens MR. Lymphoedema Functioning, Disability and Health questionnaire (Lymph-ICF): reliability and validity. Phys Ther. 2011 Jun;91(6):944-57. doi: 10.2522/ptj.20100087. Epub 2011 Apr 14. PMID 21493748
- [Background] Devoogdt N, Lemkens H, Geraerts I, Van Nuland I, Flour M, Coremans T, Christiaens MR, Van Kampen M. A new device to measure upper limb circumferences: validity and reliability. Int Angiol. 2010 Oct;29(5):401-7. PMID 20924341
- [Background] Devoogdt N, Pans S, De Groef A, Geraerts I, Christiaens MR, Neven P, Vergote I, Van Kampen M. Postoperative evolution of thickness and echogenicity of cutis and subcutis of patients with and without breast cancer-related lymphedema. Lymphat Res Biol. 2014 Mar;12(1):23-31. doi: 10.1089/lrb.2013.0028. Epub 2014 Feb 6. PMID 24502300
- [Background] Gebruers N, Truijen S, Engelborghs S, De Deyn PP. Volumetric evaluation of upper extremities in 250 healthy persons. Clin Physiol Funct Imaging. 2007 Jan;27(1):17-22. doi: 10.1111/j.1475-097X.2007.00708.x. PMID 17204033
- [Background] Tan IC, Maus EA, Rasmussen JC, Marshall MV, Adams KE, Fife CE, Smith LA, Chan W, Sevick-Muraca EM. Assessment of lymphatic contractile function after manual lymphatic drainage using near-infrared fluorescence imaging. Arch Phys Med Rehabil. 2011 May;92(5):756-764.e1. doi: 10.1016/j.apmr.2010.12.027. PMID 21530723
- [Derived] De Vrieze T, Gebruers N, Nevelsteen I, Thomis S, De Groef A, Tjalma WAA, Belgrado JP, Vandermeeren L, Monten C, Hanssens M, Asnong A, Dams L, Van der Gucht E, Heroes AK, Devoogdt N. Does Manual Lymphatic Drainage Add Value in Reducing Suprafascial Fluid Accumulation and Skin Elasticity in Patients With Breast Cancer-Related Lymphedema? Phys Ther. 2022 Dec 6;102(12):pzac137. doi: 10.1093/ptj/pzac137. PMID 36209432
- [Derived] De Vrieze T, Gebruers N, Nevelsteen I, Fieuws S, Thomis S, De Groef A, Tjalma WA, Belgrado JP, Vandermeeren L, Monten C, Hanssens M, Devoogdt N. Manual lymphatic drainage with or without fluoroscopy guidance did not substantially improve the effect of decongestive lymphatic therapy in people with breast cancer-related lymphoedema (EFforT-BCRL trial): a multicentre randomised trial. J Physiother. 2022 Apr;68(2):110-122. doi: 10.1016/j.jphys.2022.03.010. Epub 2022 Apr 12. PMID 35428594
- [Derived] Thomis S, Helberg M, Kleiman J, Vrieze T, Heroes AK, Fourneau I, Devoogdt N. The Interrater Reliability of the Scoring of the Lymphatic Architecture and Transport Through Near-InfraRed Fluorescence Lymphatic Imaging in Patients with Breast Cancer-Related Lymphedema. Lymphat Res Biol. 2022 Apr;20(2):133-143. doi: 10.1089/lrb.2020.0105. Epub 2021 Jun 2. PMID 34077678
- [Derived] De Vrieze T, Gebruers N, Nevelsteen I, Tjalma WAA, Thomis S, De Groef A, Dams L, Haenen V, Devoogdt N. Breast cancer-related lymphedema and its treatment: how big is the financial impact? Support Care Cancer. 2021 Jul;29(7):3801-3813. doi: 10.1007/s00520-020-05890-3. Epub 2020 Nov 24. PMID 33236211
- [Derived] Thomis S, Dams L, Fourneau I, De Vrieze T, Nevelsteen I, Neven P, Gebruers N, Devoogdt N. Correlation Between Clinical Assessment and Lymphofluoroscopy in Patients with Breast Cancer-Related Lymphedema: A Study of Concurrent Validity. Lymphat Res Biol. 2020 Dec;18(6):539-548. doi: 10.1089/lrb.2019.0090. Epub 2020 Mar 25. PMID 32208953
- [Derived] De Vrieze T, Gebruers N, Nevelsteen I, Tjalma WAA, Thomis S, De Groef A, Dams L, Van der Gucht E, Devoogdt N. Physical activity level and age contribute to functioning problems in patients with breast cancer-related lymphedema: a multicentre cross-sectional study. Support Care Cancer. 2020 Dec;28(12):5717-5731. doi: 10.1007/s00520-020-05375-3. Epub 2020 Mar 19. PMID 32193692
- [Derived] De Vrieze T, Frippiat J, Deltombe T, Gebruers N, Tjalma WAA, Nevelsteen I, Thomis S, Vandermeeren L, Belgrado JP, De Groef A, Devoogdt N. Cross-cultural validation of the French version of the Lymphedema Functioning, Disability and Health Questionnaire for Upper Limb Lymphedema (Lymph-ICF-UL). Disabil Rehabil. 2021 Sep;43(19):2797-2804. doi: 10.1080/09638288.2020.1716271. Epub 2020 Jan 28. PMID 31990592
- [Derived] De Vrieze T, Gebruers N, Nevelsteen I, Tjalma WAA, Thomis S, De Groef A, Dams L, Devoogdt N. Responsiveness of the Lymphedema Functioning, Disability, and Health Questionnaire for Upper Limb Lymphedema in Patients with Breast Cancer-Related Lymphedema. Lymphat Res Biol. 2020 Aug;18(4):365-373. doi: 10.1089/lrb.2019.0073. Epub 2020 Jan 22. PMID 31971890
- [Derived] De Vrieze T, Nevelsteen I, Thomis S, De Groef A, Tjalma WAA, Gebruers N, Devoogdt N. What are the economic burden and costs associated with the treatment of breast cancer-related lymphoedema? A systematic review. Support Care Cancer. 2020 Feb;28(2):439-449. doi: 10.1007/s00520-019-05101-8. Epub 2019 Oct 28. PMID 31656987
- [Derived] De Vrieze T, Gebruers N, Nevelsteen I, De Groef A, Tjalma WAA, Thomis S, Dams L, Van der Gucht E, Penen F, Devoogdt N. Reliability of the MoistureMeterD Compact Device and the Pitting Test to Evaluate Local Tissue Water in Subjects with Breast Cancer-Related Lymphedema. Lymphat Res Biol. 2020 Apr;18(2):116-128. doi: 10.1089/lrb.2019.0013. Epub 2019 Jul 19. PMID 31329510
- [Derived] De Vrieze T, Vos L, Gebruers N, De Groef A, Dams L, Van der Gucht E, Nevelsteen I, Devoogdt N. Revision of the Lymphedema Functioning, Disability and Health Questionnaire for Upper Limb Lymphedema (Lymph-ICF-UL): Reliability and Validity. Lymphat Res Biol. 2019 Jun;17(3):347-355. doi: 10.1089/lrb.2018.0025. Epub 2019 Feb 12. PMID 30759059

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Started | 65 | 64 | 65
Post Intensive Treatment Phase (= Primary Endpoint) | 63 | 63 | 64
Completed | 60 (post follow-up phase) | 61 (post follow-up phase) | 61 (post follow-up phase)
Not Completed | 5 | 3 | 4
Not completed — Death | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 3
Not completed — Illness | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD | Total
Number analyzed (Participants) | 65 | 64 | 65 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10.8) | 62 (9.5) | 61 (9.0) | 61 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 63 | 65 | 193
  Male | 0 | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 65 | 64 | 65 | 194
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 27.6 (5) | 28.8 (5.6) | 27.8 (6.1) | 28.1 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Lymphoedema Volume at the Level of the Arm/ Hand
Description: = the ratio at the different time points; The (inter-limb) ratio = Relative excessive lymphoedema volume of the arm/ hand = [(volume arm + volume hand affected side) / (corrected volume arm + corrected volume hand healthy side)]; Volume arm is determined by performing circumference measurements and calculating the volume with the formula of the truncated cone; Volume hand is determined by the water displacement method; The volume of the non-dominant hand/arm is on average 3.3% smaller than the dominant hand/arm, therefore is the volume of the arm at the healthy side corrected for hand dominance
Time Frame: Primary endpoint = After 3 weeks of intensive treatment
Population: At the post-intensive assessment, 5 patients dropped-out of which 4 patients (2%) were lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: Inter-limb ratio
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 65 | 64 | 65
Inter-limb ratio
  Baseline | 1.228 [1.190 to 1.266] | 1.249 [1.211 to 1.288] | 1.218 [1.181 to 1.256]
  Post intensive treatment phase: number analyzed (Participants) | 63 | 63 | 64
  Post intensive treatment phase | 1.175 [1.144 to 1.207] | 1.197 [1.165 to 1.229] | 1.164 [1.133 to 1.195]

2. Primary Outcome: Stagnation of Fluid at Level of the Shoulder/ Trunk
Description: Ratio PWC% at the different time intervals
  = PWC% affected side / PWC% healthy side Measured with the MoistureMeterD compact at the level of shoulder and trunk where after a mean ratio PWC% is calculated
Time Frame: Primary endpoint = After 3 weeks of intensive treatment
Population: At the post-intensive assessment, 5 patients dropped-out of which 4 patients (2%) were lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: Inter-limb ratio
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 65 | 64 | 65
Inter-limb ratio
  Baseline | 1.045 [1.024 to 1.065] | 1.051 [1.030 to 1.072] | 1.057 [1.036 to 1.078]
  Post intensive phase: number analyzed (Participants) | 63 | 63 | 64
  Post intensive phase | 1.088 [1.069 to 1.108] | 1.059 [1.040 to 1.077] | 1.077 [1.058 to 1.096]

3. Secondary Outcome: Extracellular Fluid in the Upper Limb
Description: L-Dex score, measured with Impedimed BIS device at the different time points Amount of extracellular fluid = represented by L-Dex score This outcome is calculated and displayed on the Impedimed BIS device, and represents the difference in the amount of extracellular fluid in the affected upper limb compared to the unaffected upper limb. Normal L-Dex scores range between -10 and +10. A score outside this range, represents lymphedema. A higher number, represents a worse score.
Time Frame: After 3 weeks of intensive treatment, 1, 3, 6 months of maintenance treatment and 6 months of follow-up
Population: At the post-intensive assessment, 5 patients dropped-out of which 4 patients (2%) were lost to follow-up. At the end of the maintenance phase (P6), only 3 additional patients (1.5%) were lost to follow-up. At the end of the follow-up phase (P12), one additional patient was lost to follow-up (12 patients in total since baseline or 6%).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 65 | 64 | 65
score on a scale
  Baseline | 33.1 [26.1 to 40.1] | 32.3 [25.3 to 39.3] | 34.9 [28 to 41.8]
  Post-intensive: number analyzed (Participants) | 63 | 63 | 64
  Post-intensive | 24.4 [19.1 to 29.6] | 25.4 [20.2 to 30.7] | 23.9 [18.7 to 29.1]
  1M maintenance: number analyzed (Participants) | 63 | 63 | 64
  1M maintenance | 30 [22.2 to 37.8] | 29.5 [21.6 to 37.3] | 25.3 [17.6 to 33]
  3M maintenance: number analyzed (Participants) | 61 | 63 | 63
  3M maintenance | 20.9 [17.1 to 28.5] | 22.2 [17.8 to 26.5] | 21.1 [16.8 to 25.4]
  6M maintenance: number analyzed (Participants) | 62 | 62 | 63
  6M maintenance | 22.8 [17.1 to 28.5] | 22.6 [16.8 to 28.3] | 21.6 [16 to 27.3]
  6M follow-up: number analyzed (Participants) | 60 | 61 | 61
  6M follow-up | 28.1 [20 to 36.2] | 24.1 [16 to 32.3] | 25.4 [17.3 to 33.4]

4. Secondary Outcome: Thickness of Cutis and Subcutis of Arm and Trunk Measured With Ultrasound
Description: Analyses for change in thickness of cutis + subcutis were performed:
  Relative excessive thickness of the cutis+subcutis (inter-limb ratio of cutis+subcutis in mm) = Thickness of cutis+subcutis (mm) affected side / thickness of cutis+subcutis (mm) healthy side Arm: Reference points 1, 2, 3, 5, 6, 7 where after a mean ratio thickness of cutis+subcutis is calculated
Time Frame: After 3 weeks of intensive treatment and 6 months of maintenance treatment and 6 months of follow-up
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Inter-limb ratio
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 65 | 64 | 65
Inter-limb ratio
  Baseline | 1.52 [1.42 to 1.63] | 1.44 [1.34 to 1.55] | 1.45 [1.35 to 1.56]
  Post-intensive: number analyzed (Participants) | 63 | 63 | 64
  Post-intensive | 1.36 [1.27 to 1.47] | 1.38 [1.30 to 1.47] | 1.36 [1.28 to 1.45]
  6M maintenance: number analyzed (Participants) | 62 | 62 | 63
  6M maintenance | 1.35 [1.27 to 1.44] | 1.40 [1.31 to 1.49] | 1.29 [1.21 to 1.37]
  6M follow-up: number analyzed (Participants) | 60 | 61 | 61
  6M follow-up | 1.31 [1.22 to 1.41] | 1.40 [1.30 to 1.51] | 1.34 [1.24 to 1.44]

5. Secondary Outcome: Problems in Functioning Related to Development of Breast Cancer-related Lymphoedema
Description: Different scores are obtained from the questionnaire. Each of the 29 questions has to be scored on a 11-point Likert scale between 0 and 10 (instead of a VAS between 0 and 100). The total score of the Lymph-ICF-UL is equal to the sum of the scores on the questions divided by the total number of answered questions and multiplied by 10. In addition, a score is determined for each of the five domains of the Lymph-ICFUL: (1) physical function, (2) mental function, (3) household activities, (4) mobility activities, and (5) life and social activities.
  Thus, the total score on the Lymph-ICF-UL and the score on the five domains range between 0 and 100. The higher the score, the more problems in functioning.
Time Frame: After 3 weeks of intensive treatment, 1, 3, 6 months of maintenance treatment and 6 months of follow-up
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 65 | 64 | 65
score on a scale
  Baseline | 38.0 [32.9 to 43.1] | 35.7 [30.6 to 40.8] | 38.1 [33.0 to 43.1]
  Post-intensive: number analyzed (Participants) | 63 | 63 | 64
  Post-intensive | 29.0 [24.3 to 33.6] | 27.7 [23.0 to 32.4] | 32.1 [27.5 to 36.7]
  1M maintenance: number analyzed (Participants) | 63 | 63 | 64
  1M maintenance | 27.8 [23.3 to 32.3] | 24.6 [20 to 29.1] | 28.8 [24.3 to 33.3]
  3M maintenance: number analyzed (Participants) | 61 | 63 | 63
  3M maintenance | 23.3 [18.8 to 27.8] | 25.4 [20.8 to 29.9] | 25.2 [20.7 to 29.8]
  6M maintenance: number analyzed (Participants) | 62 | 62 | 63
  6M maintenance | 25.3 [20.5 to 30] | 24.5 [19.7 to 29.3] | 27.5 [22.8 to 32.3]
  6M follow-up: number analyzed (Participants) | 60 | 61 | 61
  6M follow-up | 23.2 [18.5 to 27.9] | 24.2 [19.5 to 28.9] | 26 [21.3 to 30.7]

6. Secondary Outcome: Elasticity of Skin and Subcutaneous Tissue of Arm and Trunk Using the SkinFibrometer
Description: Induration force is presented in Newton (N) by the device. Relative difference in skin elasticity (induration force inter-limb ratio) = Skin elasticity affected side / skin elasticity healthy side Arm: Reference points 1, 2, 3, 5, 6, 7 where after a mean induration ratio is calculated
Time Frame: After 3 weeks of intensive treatment, 1, 3, 6 months of maintenance treatment and 6 months of follow-up
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Inter-limb ratio
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 65 | 64 | 65
Inter-limb ratio
  Baseline | 1.28 [1.19 to 1.37] | 1.26 [1.17 to 1.35] | 1.41 [1.31 to 1.51]
  Post-intensive treatment: number analyzed (Participants) | 63 | 63 | 64
  Post-intensive treatment | 1.11 [1.04 to 1.18] | 1.06 [1 to 1.13] | 1.14 [1.07 to 1.21]
  1M maintenance: number analyzed (Participants) | 63 | 63 | 64
  1M maintenance | 1.15 [1.08 to 1.23] | 1.07 [1.01 to 1.14] | 1.15 [1.11 to 1.26]
  3M maintenance: number analyzed (Participants) | 61 | 63 | 63
  3M maintenance | 1.16 [1.10 to 1.23] | 1.07 [1.01 to 1.14] | 1.15 [1.08 to 1.22]
  6M maintenance: number analyzed (Participants) | 62 | 62 | 63
  6M maintenance | 1.13 [1.07 to 1.20] | 1.10 [1.04 to 1.17] | 1.14 [1.08 to 1.22]
  6M follow-up: number analyzed (Participants) | 60 | 61 | 61
  6M follow-up | 1.19 [1.11 to 1.27] | 1.07 [1.01 to 1.14] | 1.15 [1.08 to 1.23]

7. Secondary Outcome: Quality of Life Score
Description: At the end of each assessment, subjects are asked to fill in the questionnaire individually Questionnaire counts 16 + 1 questions, which relate to the following 5 domains: physical symptoms; physical wellbeing, psychological symptoms; existential wellbeing and support A Likert scale with 11 possibilities (0-10) is used for the 16 questions and part D is an open question Each question corresponds to a score between 0 (very bad) and 10 (excellent); a total score and 5 different domain scores are calculated (each between 0 and 10) A lower score indicates a lower Quality of Life
Time Frame: After 3 weeks of intensive treatment and 1, 3, 6 months of maintenance treatment and 6 months of follow-up
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 65 | 64 | 65
score on a scale
  Baseline | 5.96 [5.58 to 6.35] | 6.15 [5.75 to 6.54] | 5.87 [5.48 to 6.26]
  Post-intensive: number analyzed (Participants) | 63 | 63 | 64
  Post-intensive | 6.06 [5.56 to 6.46] | 6.18 [5.77 to 6.59] | 5.82 [5.41 to 6.22]
  1M maintenance: number analyzed (Participants) | 63 | 63 | 64
  1M maintenance | 6.14 [5.71 to 6.58] | 6.21 [5.77 to 6.65] | 5.98 [5.54 to 6.42]
  3M maintenance: number analyzed (Participants) | 61 | 61 | 63
  3M maintenance | 5.85 [5.38 to 6.33] | 6.10 [5.62 to 6.58] | 5.82 [5.35 to 6.30]
  6M maintenance: number analyzed (Participants) | 62 | 62 | 63
  6M maintenance | 5.92 [5.43 to 6.41] | 6.02 [5.53 to 6.52] | 6.09 [5.60 to 6.58]
  6M follow-up: number analyzed (Participants) | 60 | 61 | 61
  6M follow-up | 5.96 [5.45 to 6.47] | 5.69 [5.18 to 6.20] | 5.81 [5.30 to 6.32]

8. Secondary Outcome: Number of Episodes of Erysipelas
Description: At each clinical evaluation, it was asked to the patient if they had had an episode of erysipelas (which is an infection) between today and the previous evaluation.
  The numbers of episodes were counted, and the causes of this episode of erysipelas were described. The numbers of episodes were compared between the groups.
Time Frame: Between baseline and the end of the follow-up phase (12 months)
Population: between baseline and the end of the follow-up phase,12 patients were lost-to-follow up in total (or 6%).
Measure: Number; unit: episodes of erysipelas
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 65 | 64 | 65
episodes of erysipelas | 5 | 8 | 7

9. Secondary Outcome: Overall Treatment Satisfaction
Description: The number patients presented as a percentage that indicated that their complaints have been slightly (3), much (2) or very much improved (1) during 12 months of time
Time Frame: Between baseline and the end of the follow-up phase (12 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 60 | 61 | 61
percentage of participants | 80 | 78 | 80

10. Secondary Outcome: Manual Lymphatic Drainage (MLD)-Specific Treatment Satisfaction
Description: The mean rating of the perceived effect of the manual lymph drainage (MLD) that patients received during the study (between 0-10). The higher the score, the higher the satisfaction about the effect of the manual lymph drainage received.
Time Frame: Between baseline and the end of the follow-up phase (12 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 60 | 61 | 61
score on a scale | 8 (2) | 7 (2) | 7 (2)

11. Secondary Outcome: Local Tissue Water at the Level of the Arm and Trunk
Description: Ratio PWC% at the different time intervals
  = PWC% affected side / PWC% healthy side Measured with the MoistureMeterD compact at different measurement points where after a mean ratio PWC% is calculated Arm: Reference points 1, 2, 3, 5, 6, 7 where after a mean ratio PWC% is calculated
Time Frame: After 3 weeks of intensive treatment phase, after 1, 3, 6 months of maintenance treatments and after 6 months of follow-up
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Inter-limb ratio
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 65 | 64 | 65
Inter-limb ratio
  Baseline | 1.418 [1.365 to 1.473] | 1.354 [1.303 to 1.406] | 1.406 [1.354 to 1.459]
  Post-intensive: number analyzed (Participants) | 63 | 63 | 64
  Post-intensive | 1.372 [1.326 to 1.419] | 1.292 [1.247 to 1.336] | 1.344 [1.300 to 1.391]
  1M maintenance: number analyzed (Participants) | 63 | 63 | 64
  1M maintenance | 1.383 [1.328 to 1.438] | 1.315 [1.264 to 1.368] | 1.394 [1.340 to 1.449]
  3M maintenance: number analyzed (Participants) | 61 | 63 | 63
  3M maintenance | 1.363 [1.309 to 1.420] | 1.288 [1.236 to 1.342] | 1.358 [1.303 to 1.415]
  6M maintenance: number analyzed (Participants) | 62 | 62 | 63
  6M maintenance | 1.343 [1.290 to 1.399] | 1.298 [1.246 to 1.351] | 1.350 [1.297 to 1.405]
  6M follow-up: number analyzed (Participants) | 60 | 61 | 61
  6M follow-up | 1.343 [1.305 to 1.383] | 1.332 [1.294 to 1.373] | 1.335 [1.297 to 1.374]

12. Secondary Outcome: Thickness of the Cutis and Subcutis of the Arm and Trunk Evaluated by Palpation (Pinch Test)
Description: In total, six reference points (located at the hand (1 reference point) and arm (5 reference points)) are being evaluated and scored (0 or 1) A reference point is scored with 1 in case the skin fold thickness at the affected side is increased compared to the reference point at the non-affected side The final outcome for the arm score is the (cumulated) total score of six reference points 1, 2, 3, 5, 6, 7 (range 0-6), a higher score indicates more presence of thickened skin
Time Frame: After 3 weeks of intensive treatment, 1, 3, 6 months of maintenance treatment and 6 months of follow-up
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 65 | 64 | 65
score on a scale
  Baseline | 4.43 [4.01 to 4.85] | 4.03 [3.61 to 4.45] | 4.65 [4.23 to 5.07]
  Post-intensive: number analyzed (Participants) | 63 | 63 | 64
  Post-intensive | 4.62 [4.23 to 5] | 4.23 [3.84 to 4.63] | 4.57 [4.18 to 4.96]
  1M maintenance: number analyzed (Participants) | 63 | 63 | 64
  1M maintenance | 4.37 [3.96 to 4.78] | 4.25 [3.84 to 4.66] | 4.22 [3.81 to 4.62]
  3M maintenance: number analyzed (Participants) | 61 | 63 | 63
  3M maintenance | 4.25 [3.82 to 4.68] | 4.19 [3.76 to 4.62] | 4.22 [3.79 to 4.64]
  6M maintenance: number analyzed (Participants) | 62 | 62 | 63
  6M maintenance | 4.22 [3.77 to 4.67] | 4.03 [3.58 to 4.49] | 4.05 [3.60 to 4.50]
  6M follow-up: number analyzed (Participants) | 60 | 61 | 61
  6M follow-up | 4.09 [3.61 to 4.57] | 3.92 [3.44 to 4.40] | 4.17 [3.69 to 4.65]

13. Secondary Outcome: Hardness (Fibrosis) of the Skin at the Level of the Arm and Trunk Evaluated Through Palpation
Description: In total, six reference points (located at the hand (1 reference point) and arm (5 reference points)) are being evaluated and scored (0 or 1) A reference point is scored with 1 in case fibrosis of the skin is present The final outcome for the arm score is the (cumulated) total score of six reference points 1, 2, 3, 5, 6, 7 (range 0-6), a higher score indicates more presence of fibrosis
Time Frame: After 3 weeks of intensive treatment, 1, 3, 6 months of maintenance treatment and 6 months of follow-up
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
Number analyzed (Participants) | 65 | 64 | 65
score on a scale
  Baseline | 0.49 [0.32 to 0.67] | 0.26 [0.12 to 0.41] | 0.24 [0.10 to 0.40]
  Post-intensive: number analyzed (Participants) | 63 | 63 | 64
  Post-intensive | 0.40 [0.22 to 0.59] | 0.44 [0.26 to 0.64] | 0.56 [0.37 to 0.78]
  1M maintenance: number analyzed (Participants) | 63 | 63 | 64
  1M maintenance | 0.37 [0.21 to 0.55] | 0.52 [0.35 to 0.72] | 0.42 [0.26 to 0.61]
  3M maintenance: number analyzed (Participants) | 61 | 61 | 63
  3M maintenance | 0.17 [0.03 to 0.32] | 0.45 [0.29 to 0.64] | 0.50 [0.33 to 0.69]
  6M maintenance: number analyzed (Participants) | 62 | 62 | 63
  6M maintenance | 0.15 [0.05 to 0.25] | 0.23 [0.13 to 0.35] | 0.28 [0.17 to 0.40]
  6M follow-up: number analyzed (Participants) | 60 | 61 | 61
  6M follow-up | 0.22 [0.11 to 0.34] | 0.20 [0.09 to 0.32] | 0.24 [0.13 to 0.37]

14. Secondary Outcome: Lymphatic Architecture and Function
Description: 1. Total dermal backflow score (0-39). The higher the score, the more dermal backflow is present
  2. Amount of efferent lymphatics leaving dermal backflow areas
  3. Presence of visible lymph nodes after the break
  Raw data is currently still being analyzed in order to be able to report on the described outcome measures. At present (March 2022) these analyses are not yet performed. Therefore these results will be reported later on this year (anticipated date: July 2022).
Time Frame: After 3 weeks of intensive treatment and 6 months of maintenance treatment
Reporting Status: Not Posted, anticipated posting 2022-07

ADVERSE EVENTS:
Time Frame: Adverse events were collected between baseline and the end of the phollow-up phase (P12), which was one year post-baseline.
Description: see table (results)
Arm/Group | Fluoroscopy-guided MLD | Traditional MLD | Placebo MLD
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63 | 0/64
Other Adverse Events (participants affected / at risk) | 5/63 | 8/63 | 7/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoroscopy-guided MLD (N=63) | Traditional MLD (N=63) | Placebo MLD (N=64)
Occurence of erysipelas (not due to the trial, but due to wounds or scratches) (Blood and lymphatic system disorders) | 5 (5) | 8 (8) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT02609724/Prot_SAP_000.pdf